CLINICAL TRIAL: NCT00753142
Title: Mechanism Underlying Beta-cell Failure in Obese African Americans With History of Hyperglycemic Crises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 898-2003
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Participants with ketosis-prone diabetes (Active Comparator): Obese African Americans with type 2 diabetes with history of diabetic ketoacidosis (DKA) receiving Intralipid 20% and a glucose infusion.
  Interventions: Drug: Intralipid 20%; Drug: Glucose infusion
- Participants with ketosis-resistant diabetes (Active Comparator): Obese African American with type 2 diabetes with hyperglycemia without ketosis receiving Intralipid 20% and a glucose infusion.
  Interventions: Drug: Intralipid 20%; Drug: Glucose infusion
- Non-diabetic control group (Active Comparator): Obese African Americans without diabetes receiving a glucose infusion.
  Interventions: Drug: Glucose infusion

INTERVENTIONS:
Drug: Intralipid 20% — Participants receive a 48-hour infusion with Intralipid at 40 milliliters per hour (mL/hr).
  Arms: Participants with ketosis-prone diabetes; Participants with ketosis-resistant diabetes
Drug: Glucose infusion — Participants receive a glucose infusion consisting of 10% dextrose infused intravenously at a rate of 200 mg/m^2/min for 20 hours.

SUMMARY:
Obesity is common in African American (AA) patients with newly diagnosed diabetes who present with diabetic ketoacidosis (DKA). Despite the presentation with severe symptoms of insulinopenia and ketoacidosis, clinical and immunogenetic observations indicate that most obese AA patients with DKA have type 2 diabetes. In such patients, previous studies reveal that: a) at presentation, obese AA patients with DKA have markedly decreased pancreatic insulin secretion, lower than in obese non-DKA patients admitted with comparable hyperglycemia, but significantly greater than in lean patients with DKA; b) aggressive diabetic management results in significant improvement in beta-cell function and insulin sensitivity sufficient to allow discontinuation of insulin therapy within 3 months of follow-up. Based on these observations the researchers conclude that similar to obese patients with hyperglycemia, most obese AA with DKA have type 2 diabetes, and that although defects in both insulin secretion and insulin action are present, transient b-cell failure is the primary defect in the development of ketoacidosis.

DETAILED DESCRIPTION:
Obese AA patients with a history of DKA who later experience near-normoglycemia remission represent an ideal population in which to define the sequence of events that lead to b-cell dysfunction in type 2 diabetes. The researchers hypothesize that obese AA with DKA will prove particularly susceptible to beta-cells dysfunction due to sustained elevations of plasma glucose (glucose toxicity) and/or free fatty acid levels (lipotoxicity). This study will test beta-cell response by administering a glucose infusion to diabetic African Americans with a history of DKA, diabetic African Americans without a history of DKA, and non-diabetic African Americans.

ELIGIBILITY:
Inclusion Criteria:

* Obese African American subjects (body mass index (BMI) equal or greater than 30)
* Age 18-65
* Patients with a history of diabetic ketoacidosis as defined by the American Diabetes Association (ADA) criteria
* Patients admitted with hyperglycemia but without ketoacidosis (blood glucose greater than 400ml/dl without evidence of ketosis/ketones
* Obese nondiabetic controls (BMI >30; ruled out for diabetes with a 75g oral glucose tolerance test)

Exclusion Criteria:

* Patients with positive autoimmune markers (islet cell or glutamic acid decarboxylase (GAD) autoantibodies)
* Patients with significant medical or surgical illness, including but not limited to myocardial ischemia, congestive heart failure, chronic renal insufficiency, liver failure, and infectious processes
* Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, such as hypercortisolism, acromegaly, or hyperthyroidism
* Patients with bleeding disorders, thrombocytopenia, or abnormalities in coagulation studies
* Patients with fasting hyperglycemia (blood glucose > 120 mg/dl) after discontinuation of insulin therapy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Gosmanov AR, Smiley D, Robalino G, Siqueira JM, Peng L, Kitabchi AE, Umpierrez GE. Effects of intravenous glucose load on insulin secretion in patients with ketosis-prone diabetes during near-normoglycemia remission. Diabetes Care. 2010 Apr;33(4):854-60. doi: 10.2337/dc09-1687. Epub 2010 Jan 12. PMID 20067967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began in March 2004 and all study follow-up was completed in December 2009. The study was conducted at the Clinical Research Center at Grady Memorial Hospital in Atlanta, Georgia.
Groups:
- Ketosis-prone Diabetics: Obese African Americans with type 2 diabetes and a history of diabetic ketoacidosis (DKA) receiving a 48-hour infusion of Intralipid 20% at 40 mL/hour and a glucose infusion of 10% dextrose infused at a rate of 200 mg/m^2/min for 20 hours.
- Ketosis-resistant Diabetics: Obese African Americans with type 2 diabetes with hyperglycemia without ketosis receiving a 48-hour infusion of Intralipid 20% at 40 mL/hour and a glucose infusion of 10% dextrose infused at a rate of 200 mg/m^2/min for 20 hours.
- Non-diabetic Control Group: Obese African Americans without diabetes receiving a glucose infusion of 10% dextrose infused at a rate of 200 mg/m^2/min for 20 hours.
Period: Overall Study
Arm/Group | Ketosis-prone Diabetics | Ketosis-resistant Diabetics | Non-diabetic Control Group
Started | 8 | 7 | 13
Completed | 8 | 7 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketosis-prone Diabetics | Ketosis-resistant Diabetics | Non-diabetic Control Group | Total
Number analyzed (Participants) | 8 | 7 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (10.6) | 49.7 (8.1) | 40 (9.3) | 44 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 12 | 16
  Male | 6 | 5 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 13 | 28
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: First-Phase Insulin Release (FPIR)
Description: An arginine stimulation test was used to evaluate beta-cell function and insulin secretion. Increased glucose in the blood causes insulin to be released, beginning with a spike in insulin in the first 10 minutes and plateauing 2 to 3 later. Diminished first-phase insulin release is an early indicator of beta-cell dysfunction. Two sequential arginine stimulation tests were performed, the first set before and the second after completion of the 20-hour dextrose infusion. The first-phase insulin release (FPIR) was calculated as the sum of the insulin levels at 2, 3, 4, and 5 minutes after the arginine infusion. FPIR is expected to rise after the dextrose (glucose) infusion and FPIR generally rises less in persons with impaired glucose tolerance.
Time Frame: Hour 0, Hour 20
Measure: Mean (Standard Deviation); unit: microunits/ml
Arm/Group | Ketosis-prone Diabetics | Ketosis-resistant Diabetics | Non-diabetic Control Group
Number analyzed (Participants) | 8 | 7 | 13
microunits/ml
  Before glucose infusion | 264 (80) | 339 (221) | 197 (33)
  After glucose infusion | 359 (42) | 381 (147) | 299 (30)

2. Secondary Outcome: Number of Participants With Beta-cell Failure
Description: Pancreatic beta-cells can adapt to insulin resistance during the early stages of diabetes but continuous exposure of beta-cells to prolonged hyperglycemia can cause irreversible damage due to glucotoxicity. This study aimed to evaluate whether hyperglycemia-induced reduced beta-cell failure was the result of beta-cell exhaustion or beta-cell desensitization, however, no participants experienced beta-cell failure so this original analysis could not be performed.
Time Frame: Hour 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ketosis-prone Diabetics | Ketosis-resistant Diabetics | Non-diabetic Control Group
Number analyzed (Participants) | 8 | 7 | 13
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ketosis-prone Diabetics | Ketosis-resistant Diabetics | Non-diabetic Control Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 1/8 | 1/7 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketosis-prone Diabetics (N=8) | Ketosis-resistant Diabetics (N=7) | Non-diabetic Control Group (N=13)
hyperglycemia (Endocrine disorders) | 1 | 1 | 0 — blood sugar intermittently > 300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No